CLINICAL TRIAL: NCT05092802
Title: An Open-label, Multicenter Phase II Clinical Study to Evaluate Safety, Efficacy and PK of HLX208 for Refractory Primary Brain Tumors With BRAF Mutation
Brief Title: The Efficacy of HLX208 (BRAF V600E Inhibitor) for Refractory Primary Brain Tumors With BRAF Mutation After First-line Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX208-BT201
Record Dates: First submitted 2021-09-18; First posted 2021-10-26 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-09

CONDITIONS: Brain Tumor, Primary
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX208 (Experimental)
  Interventions: Drug: HLX208

INTERVENTIONS:
Drug: HLX208 — 450mg bid po

SUMMARY:
An open-label, multicenter phase II clinical study to evaluate safety, efficacy and PK of HLX208 for refractory primary brain tumors with BRAF mutation

ELIGIBILITY:
Inclusion Criteria:

* Age>=18Y
* Good Organ Function
* Expected survival time ≥ 3 months
* Refractory primary brain tumors with BRAF mutation that have been diagnosed
* Unable to receive surgery/radiotherapy, or have treatment failed after surgery/radiotherapy
* ECOG score 0-1;

Exclusion Criteria:

* Previous treatment with BRAF inhibitors or MEK inhibitors
* A history of other malignancies within two years, except for cured cervical carcinoma in situ, basal cell carcinoma of the skin, adenocarcinoma in situ of the lung, or tumors that do not require interventional treatment after radical surgery
* Severe active infections requiring systemic anti-infective therapy
* Other anti-tumor treatments, such as chemotherapy, targeted therapy, or radiation therapy (except palliative radiation therapy), may be given during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
ORR | from first dose to the last patient was followed up for 6 month
  Objective response rate(assessed by independent radiological review committee (IRRC) based on the RANO

SECONDARY OUTCOMES:
PFS | from the first dose until firstly confirmed and recorded disease progression or death (whichever occurs earlier)，an average of about 1 year
  Progression-free survival(PFS):assessed by IRRC and the investigator based on the RANO
DOR | from the first occurrence of a documented CR or PR (whichever recorded earlier) to the time of first documented disease progression or death (whichever occurs first)，an average of about 1 year
  Duration of response
OS | from the first dose to the time of death due to any cause，an average of about 2 year
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Cancer Hospital Affiliated to Shandong first medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No